CLINICAL TRIAL: NCT07012980
Title: Efficacy and Safety of Glofitamab, Polatuzumab Vedotin and Zanubrutinib in the First-line Treatment of Elderly Patients With Diffuse Large B-cell Lymphoma (DLBCL): A Single-center, Single-arm, Prospective, Phase II Trial
Brief Title: Glofitamab, Polatuzumab Vedotin and Zanubrutinib in First-line Elderly DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry); BeiGene (Industry)
Responsible Party: Principal Investigator, Peng Liu, Professor, Chief Physician, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHZS-DLBCL004
Record Dates: First submitted 2025-05-24; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: glofitamab; polatuzumab vedotin; zanubrutinib; first-line; elderly; frail
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab; polatuzumab vedotin; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glofitamab, polatuzumab vedotin and zanubrutinib (Experimental): Glofitamab will be administered i.v. on a step-up dosing schedule starting on Day 8 of Cycle 1 (2.5 mg), Day 15 of Cycle 1 (10 mg), followed by 30 mg on Day 1 of Cycles 2-6, with each cycle being 21 days.
  A single dose of obinutuzumab 1000 mg will be administered intravenously on Day 1 of Cycle 1.
  Polatuzumab vedotin (1.8 mg/kg) will be administered intravenously on Day 2 of Cycle 1 and on Day 1 of the subsequent Cycle 2-6 (each Q3W).
  Zanubrutinib (160mg bid p.o.) will be administered for 7 days as pretreatment and from D1 to D21 through all 12 cycles Q3W.
  Interventions: Drug: Glofitamab; Drug: Polatuzumab Vedotin; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Glofitamab — Glofitamab will be administered i.v. on a step-up dosing schedule starting on Day 8 of Cycle 1 (2.5 mg), Day 15 of Cycle 1 (10 mg), followed by 30 mg on Day 1 of Cycles 2-6, with each cycle being 21 days. A single dose of obinutuzumab 1000 mg will be administered intravenously on Day 1 of Cycle 1.
Drug: Polatuzumab Vedotin — Polatuzumab vedotin (1.8 mg/kg) will be administered intravenously on Day 2 of Cycle 1 and on Day 1 of the subsequent Cycle 2-6 (each Q3W).
  Other Names: Polivy
Drug: Zanubrutinib — Zanubrutinib (160mg bid p.o.) will be administered for 7 days as pretreatment and from D1 to D21 through all 12 cycles Q3W.

SUMMARY:
This study aims to assess the efficacy and safety of the chemotherapy-light combination of glofitamab, polatuzumab vedotin and zanubrutinib (GPZ) in elderly patients with previously untreated diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This study is a prospective, single-center, interventional, phase 2 study. Each patient screend eligible for this study will receive a combination therapy of glofitamab, zanubrutinib and polatuzumab vedotin.

ELIGIBILITY:
Inclusion Criteria:

Subjects will only be included in the study if they meet all the following criteria:

1. Written informed consent.
2. Aged 70 years old or above.
3. ECOG performance status of 0-3.
4. Histologically confirmed CD20 positive DLBCL.
5. At least one measurable site of disease.
6. Patient did not receive any prior lymphoma therapy.
7. Patient has a life expectancy (in the opinion of the investigator) of at least 12 weeks.
8. Patient has adequate liver function:

   * Total bilirubin ≤1.5 x ULN (≤3 x ULN in patients with Gilbert's syndrome).
   * AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤3 x ULN. o Patients with documented liver involvement: AST and/or ALT ≤5 x ULN.
9. Patient as adequate hematological function, unless due to lymphoma:

   * Hemoglobin ≥9.0 g/dL within 7 days before the first treatment.
   * Absolute neutrophil count of ≥1.0 x 109 cells/L (1,000/μL).
   * Platelet count of ≥75 x 109 cells/L (75,000/μL). Note: Transfusion of RBCs and platelets is allowed to reach the inclusion criteria. In case screening procedures are leading to situations that would exclude the patient from study participation (such as Hb value below entry criteria), the patient may still be enrolled into the trial after consultation with the principal investigator.
10. Patient has adequate renal function:

    * Creatinine ≤ 1.5 x ULN, or
    * Creatinine clearance (CrCl) calculated by Cockcroft-Gault formula of ≥ 30 mL/min for patients in whom, in the Investigator's judgment, serum creatinine levels do not adequately reflect renal function.

Exclusion Criteria:

Subjects will not be included in the study if any of the following criteria apply:

1. History of severe cardiac disease: New York Heart Association (NYHA) grade 3-4, congestive heart failure, myocardial infarction or cerebrovascular accident within the past 3 months, unstable arrhythmias, or unstable angina or history of multiple cardiovascular events) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).

   Note: Congestive heart failure NYHA II patients can be included if they provide an LVEF >40%.;
2. Patient with current or history of CNS lymphoma.
3. Patient with uncontrolled severe infection, whether bacterial (e.g., tuberculosis), viral (including, but not limited to severe pneumonia, COVID-19, Epstein-Barr virus [EBV], cytomegalovirus [CMV], hepatitis B, hepatitis C, and HIV], fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks prior to study enrollment.

   Note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
4. Patient with current > Grade 1 peripheral neuropathy.
5. Any other prior malignancy than non-melanoma skin cancer or stage 0 (in situ) cervical carcinoma, unless treated with curative intent, and without relapse since 2 years, or low grade prostate cancer, not in need of treatment
6. Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study.
7. Known hypersensitivity to Chinese hamster ovary (CHO) cell products or to any component of the zanubrutinib, polatuzumab vedotin, obinutuzumab, or glofitamab and/or to the contrast agents used in the study.

   -

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) rate | From the day of inclusion until disease progression (PD) or relapse after complete remission (CR) as per Lugano Classification of 2014, or death due to any cause, whichever occurs first, assessed up to 39 months.
  defined as the time from the day of inclusion until disease progression (PD) or relapse after complete remission (CR) as per Lugano Classification of 2014, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
CR rate | up to 12 cycles, an avergae of 11 months
  defined as the number of patients achieving CR divided by the number of analyzable patients.
DoR | From documentation of CR/PR until relapse/progression or death due to any reason without documented relapse. Assessed up to 39 months.
  defined as the time from documentation of CR/PR until relapse/progression or death due to any reason without documented relapse. Patients who have not experienced an event at the time of analysis will be censored at the most recent date of disease assess
Incidence of treatment-related death rate | defined as the number of treatment related deaths during therapy or up to 2 months after the end of study treatment, but before the start of further treatment, divided by the number of analyzable patients.
  defined as the number of treatment related deaths during therapy or up to 2 months after the end of study treatment, but before the start of further treatment, divided by the number of analyzable patients.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: IPD could be requested by contacting the corresponding author via email after publication.